CLINICAL TRIAL: NCT02074865
Title: Children's Antibiotic Resistant Infections in Low Income Countries
Acronym: ChARLI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut Pasteur in Madagascar (subject recruitment) (Unknown); department of International cooperation of Monaco (funding) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2012-11 ChARLI
Record Dates: First submitted 2013-07-10; First posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At birth, for therapeutic management of the newborns in the presence of a risk factor for infection :gastric fluid, external auditory canal swabs, anal swabs, placental biopsy. Before empirical antibiotic treatment: blood cultures, blood sampling for CRP determination.In the presence of particular warning signs of infection chest X ray and lumbar puncture.
  During the follow-up, for therapeutic management of the newborns if the child has a suspected infection : urine samples, blood for blood cultures and Blood formula and C-reactive protein (CRP) detrmination; rhinopharyngeal fluid samples, lumbar puncture in febrile children under the age of three months; and thick blood smears if the child has a fever.
  Samples based on the presence of particular warning signs of infection: stool samples, eye or ear swabbing, chest X
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- newborns
  Interventions: Biological: biological samples

INTERVENTIONS:
Biological: biological samples

SUMMARY:
The main challenge of the ChARLI program is to assess the clinical burden of severe neonatal and childhood bacterial infections in low-income countries,in particular those caused by antibiotic resistant bacteria. This program will address both healthcare associated, as well as community acquired infections. Beside its main challenge, the ChARLI program will also allow the assessment of the economic burden of these infections, the improvement of their medical care and then ultimately help to set public health interventions and guide public health measures necessary to combat bacterial infections and bacterial resistance in children. It will also lead to set up more basic research investigation to better understand how pathogenic and epidemic may be the resistant clones in these countries and to experiment innovative strategies devoted to prevent these infections.

In order to achieve these objectives, an international paediatric cohort will be created, and monitored a platform. This will be done first within the Institut Pasteur International Network (IPIN) and possibly extended in some others low income countries where the IPIN has no center. This constituted initiative will represent the first international pediatric program of its size to be located in low-income countries and specifically focusing severe bacterial infections and bacterial resistance to antibiotics

ELIGIBILITY:
Inclusion Criteria:

* Neonate born to parents living in the study zone of a participating country
* Parents of the neonate not intending to move away from the study zone during the follow-up period
* Legal guardians of the neonate informed about the way in which the study is to be carried out and about the collection of biological samples
* Legal guardians of the neonate having no objection to the collection of biological samples
* Authorisation from at least one of the legal guardians of the child, in the form of a signed informed consent form.

Exclusion Criteria:

* Stillborn neonate
* Parents of the neonate living outside the study zone of a participating country
* Neonate born to parents planning to move away from the study zone of a participating country during the follow-up period
* At least one of the legal guardians of the neonate not informed about the study or about the collection of biological samples
* At least one of the legal guardians of the neonate opposed to the collection of biological samples.
* Neonate already participating in another biomedical study.

Ages: 1 Minute to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: newborns
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of infections with bacteria resistant to antibiotics in neonates and young children (up to 18 months of age). | 27 months

SECONDARY OUTCOMES:
Bacterial aetiology of neonatal infection in low income countries and its resistance | 27 months
Identification of factors responsible of the dissemination and transmission of multiresistant resistant bacteria in low incomes countries | 27 months

CONTACTS AND LOCATIONS:
Locations (1):
- institut pasteur in Madagascar, Antananarivo, Madagascar

REFERENCES:
- See also: Related Info — http://www.charliproject.org/